CLINICAL TRIAL: NCT04013243
Title: Effect of Magnesium on Maintenance Dose of Rocuronium for Deep Neuromuscular Blockade During Robotic Radical Prostatectomy
Brief Title: Effect of Magnesium on Dose of Rocuronium for Deep Neuromuscular Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, Clinical Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B-1902/523-007
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Magnesium Sulfate Causing Adverse Effects in Therapeutic Use; Neuromuscular Blockade
Keywords: Magnesium
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate group (Active Comparator): magnesium sulphate 50mg/kg in normal saline 50ml infusion for 10minutes for loading dose followed by 15mg/kg/hr for continuous infusion
  Interventions: Drug: Magnesium Sulfate
- Placebo group (Placebo Comparator): Normal Saline 50ml infusion for loading dose followed by continuous infusion for same dose of magnesium.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — magnesium sulphate 50mg/kg in normal saline 50ml infusion for 10minutes for loading dose followed by 15mg/kg/hr for continuous infusion
  Arms: Magnesium Sulfate group
Drug: Placebo — Normal Saline 50ml infusion for loading dose followed by continuous infusion for same dose of magnesium.
  Arms: Placebo group

SUMMARY:
It is well known that magnesium enhances the effect of neuromuscular blocking agents such as rocuronium. However, it is not known how much magnesium can reduce neuromuscular blocking agents in maintaining deep neuromuscular blockade. Through this study, the investigators will quantitatively analyze the rocuronium saving effect of magnesium.

DETAILED DESCRIPTION:
It is well known that magnesium potentiate the effect of neuromuscular blocking agents. It prolonged the duration of rocuronium and reduces the onset time of rocuronium. Magnesium acts on motor end plate, where magnesium reduces the release of prejunctional acetylcholine, thereby decreasing the muscle membrane excitability. However, the quantitative rocuronium saving effect of magnesium is not clear. This study's hypothesis is that magnesium would reduce the amount of rocuronium. And the investigators want to evaluate how much magnesium can reduce the amount of rocuronium. Secondary outcome is the effects of magnesium on recovery time, postoperative pain, nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective robot assisted radical prostatectomy, between 20 and 80 years with a American Society of Anesthesiologists physical status classification of I or II

Exclusion Criteria:

* Conduction abnormalities in preoperative EKG such as Atrioventricular block, sinus pause
* Glomerular filtration rate <60ml/min/1.73m2
* Allergy to rocuronium, sugammadex, magnesium
* Medications that interfered with muscle activity
* Neuromuscular disease
* Hypermagnesemia

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
rocuronium amount | perioperative - until 48hours
  total rocuronium/weight/infusion time

SECONDARY OUTCOMES:
recovery time | perioperative - until 48hours
  time from sugammadex injection to Train-of-four ratio 0.9
postoperative pain | at postoperative 30minutes, 6hours, 24hours
  11 point Numerical Rating Scale; 0 (no pain) to 10 (worst imaginable pain), rescue medication
postoperative nausea and vomiting | at postoperative 30minutes, 6hours, 24hours
  Numerical Rating Scale(0-10), rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Ah-young Oh, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Queiroz Rangel Micuci AJ, Vercosa N, Filho PAG, de Boer HD, Barbosa DD, Cavalcanti IL. Effect of pretreatment with magnesium sulphate on the duration of intense and deep neuromuscular blockade with rocuronium: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):502-508. doi: 10.1097/EJA.0000000000001003. PMID 30985540
- [Derived] Han J, Jeon YT, Ryu JH, Koo CH, Nam SW, Cho SI, Oh AY. Effects of magnesium on the dose of rocuronium for deep neuromuscular blockade: A randomised controlled trial. Eur J Anaesthesiol. 2021 Apr 1;38(4):432-437. doi: 10.1097/EJA.0000000000001329. PMID 32890015